CLINICAL TRIAL: NCT05290207
Title: A Study of Endocrine Hormone Changes in Newly Diagnosed Patients With Type 2 and Type 1 Diabetes Using Hyperinsulinaemic Hypoglycaemic Clamp Technique
Brief Title: The Different Response of Endocrine Hormones to Hypoglycemia in Patients With Type 1 or Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Jian-hua Ma, Professor, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: KY20220124-07
Record Dates: First submitted 2022-03-17; First posted 2022-03-22 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2022-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Newly diagnosed male obese patients with type 2 diabetes
  Interventions: Diagnostic Test: The hyperinsulinaemic hypoglycaemic clamp
- Newly diagnosed male non-obese patients with type 2 diabetes
  Interventions: Diagnostic Test: The hyperinsulinaemic hypoglycaemic clamp
- Newly diagnosed male patients with type 1 diabetes
  Interventions: Diagnostic Test: The hyperinsulinaemic hypoglycaemic clamp
- Healthy, non-obese men
  Interventions: Diagnostic Test: The hyperinsulinaemic hypoglycaemic clamp

INTERVENTIONS:
Diagnostic Test: The hyperinsulinaemic hypoglycaemic clamp — Glucose will be clamped at 5.0 mmol/L for approximately 30 minutes, and then be lowered to 3.0 mmol/L for 30 minutes

SUMMARY:
Endocrine hormones, not only blood glucose responsive hormones, but also sexual hormones, thyroid hormones, growth hormones and so on, may have response and activites in hypoglycemia. However, the different responses of endocrine hormones to hypoglycemia in patients With diabetes remain unclear.

DETAILED DESCRIPTION:
This study will observe the changes of insulin, C-peptide, glucagon, growth hormone, IGF-1, ACTH, cortisol, thyroid function, sexual hormone in newly diagnosed men with type 2 and type 1 diabetes mellitus using hyperinsulinaemic hypoglycaemic clamp technique

ELIGIBILITY:
Inclusion Criteria:

- Patients

* newly diagnosed male patients with type 1 or type 2 diabetes (diagnostic criteria of World Health Organization)
* aged 18-50 years
* has not been treated with any hypoglycemic drugs
* HbA1c>9% Normal subjects: healthy and had no known illness

Exclusion Criteria:

* patients with insulin allergy.
* any history of hypoglycemic agent intake or were presently taking hypoglycemic agents
* any abnormality in liver or kidney function on blood and urine investigations
* any history of systemic corticosteroid use in 3 months
* any recent infections or acute medical events
* any other obvious conditions or associated diseases determined by the researcher: such as severe cardiopulmonary diseases, endocrine diseases, neurological diseases, tumors and other diseases, other pancreatic diseases, history of mental diseases.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal subjects and newly diagnosed male patients with type 1 or type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
endocrine hormone changes | 20 minutes
  changes of endocrine hormones during hyperinsulinaemic hypoglycaemic clamps

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing Medical Univesity, Nanjing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhou Y, Zhou J, Ma J, Yan R, Yuan L, Huang R, Shen Y, Ding B. Comparative Evaluation of Responsiveness of Insulin Counter-Regulatory Hormones and Insulin Resistance to Hypoglycemia in Newly Diagnosed Type 1 Diabetes Mellitus Man. Diabetes Metab Syndr Obes. 2025 Nov 21;18:4309-4317. doi: 10.2147/DMSO.S554306. eCollection 2025. PMID 41306512